CLINICAL TRIAL: NCT01926132
Title: High-dose Ascorbic Acid Intravenous Injection Decreases Mitochondrial DNA Damage in Chronic Fatigue Patients: Randomized-controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3-2012-0154
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Fatigue
Keywords: ascorbic acid; fatigue; mitochondrial DNA; patient for more than 6 months
MeSH Terms: conditions — Fatigue | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ascorbic acid 10g/20ml (Experimental): Normal Saline 130ml+ ascorbic acid 10g/20ml , covered bottle for the blind allocation
  Interventions: Drug: ascorbic acid 10g/20ml
- Normal Saline 150ml (Active Comparator): Normal Saline 150ml, covered bottle
  Interventions: Drug: Normal Saline 150ml

INTERVENTIONS:
Drug: ascorbic acid 10g/20ml — ascorbic acid 10g/20cc intravenous injection for 40mins
  Arms: ascorbic acid 10g/20ml
Drug: Normal Saline 150ml — Normal Saline 150ml intravenous injection for 40mins
  Arms: Normal Saline 150ml

SUMMARY:
Reactive Oxygen Species (ROS) can cause oxidative damage, resulting in oxidation of lipids, proteins and DNA. In fatigue patients, there are some evidences of oxidative damage to DNA. Ascorbic acid was known to protect mitochondrial injury against oxidative stress by depolarizing the mitochondrial membrane. The copy number of mitochondrial DNA(mtDNA) was suggested mitochondrial gene stability and biogenesis and reflected mitochondrial function. There is no evidence ascorbic acid would decrease the mtDNA damage in fatigue patients. The investigators hypothesized that decreasing in mtDNA copy number in salivary and blood sample may be reversed by high-dose vitamin C intravenous injection in fatigue patients. The investigators will compare the mtDNA copy number and fatigue scale between moderate-severe fatigue patients and control group that had not malignant and chronic illness by a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with above 18 years old and 6 month fatigue duration
2. Moderate to severe fatigue scale (Brief fatigue inventory-Korean version scale ≥ 4)
3. Normal limit values in the screening test (White blood cell count, Hemoglobin, Creatinine, SGOT/SGPT, Thyroid stimulating hormone, Urinalysis)
4. Normal limit values in glucose 6 phosphate dehydrogenase level
5. Agree the subjects explanation

Exclusion Criteria:

1. pregnancy and lactation
2. acute common cold, acute gastroenteritis, uncontrolled diabetes, uncontrolled hypertension, liver disease or renal disease
3. previous medical history, affectable by high-dose ascorbic acid (gout, renal calculi and glucose 6 phosphate dehydrogenase deficiency)
4. hypersensitivity from ascorbic acid
5. vitamin supplement intake until 2 days ago
6. drug interactions with ascorbic acid ( aspirin, Fe, phenytoin, estrogen, tetracycline, coumarin, corticosteroid)
7. Do not read a consent fom

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
fatigue scale | 2 weeks after 10g ascorbic aicd intravenous injection

SECONDARY OUTCOMES:
mitochondrial DNA copy number on blood and salivary samples | 2 weeks after 10g ascorbic aicd intravenous injection

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, Seoul, South Korea